CLINICAL TRIAL: NCT01673490
Title: A Pivotal, Open-label Trial Assessing the Safety and Efficacy of the 0.5 mg Dutasteride and 0.4 mg Tamsulosin Combination Once Daily for Six Months in Patients With Benign Prostatic Hyperplasia
Brief Title: Safety and Efficacy of 0.5mg Dutasteride and 0.4mg Tamsulosin Combination Once Daily for Six Months for Benign Prostatic Hyperplasia
Acronym: FDC114785
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sole investigative site refused to accept the amended protocol and declined to continue the study. There was no safety signal nor any other reason.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114785
Record Dates: First submitted 2012-06-28; First posted 2012-08-28 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; dutasteride and tamsulosin
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combodart/Duodart (Experimental): Single arm testing the efficacy/safety of the combinnation of Dutasteride/Tamsulosin
  Interventions: Drug: Dutasteride/Tamsulosin

INTERVENTIONS:
Drug: Dutasteride/Tamsulosin — 0.5 mg dutasteride/ 0.4 mg tamsulosin once daily for the duration of 180 day -treatment
  Other Names: Duodart; combodart

SUMMARY:
Open-label, 6 month-treatment with the IP in all subjects. - Sample size: A total of 90 subjects will be enrolled so that among them at least 57 will complete the 6-month treatment period and evaluable for analysis.

-Primary objective: To assess the safety of 0.5 mg dutasteride/0.4 mg tamsulosin combination therapy for six month in BPH patients by monitoring category, frequency and severity of adverse events encountered during the treatment period.

-Secondary objective: To assess the efficacy of 0.5 mg dutasteride/0.4 mg tamsulosin combination therapy with regard to symptom improvement in BPH patients by monitoring and analyzing of changes in IPSS and Qmax after 6 months of treatment.

DETAILED DESCRIPTION:
Visit 0 or Screening Visit (M0) - D0 + 2): Following tasks will be performed: ICF collection, subject code assignment, physical examination (vital signs, demographic data, medical history); checking of inclusion and exclusion criteria: prostate symptom score according to IPSS, laboratory tests (hematology, blood chemistry, electrolytes, total PSA level, free-to-total PSA ratio, Qmax, urinalysis, transrectal prostate ultrasonography (TRUS), 12-lead electrocardiography (ECG), scoring of Sexual Function Questionnaire (SFQ), concomitant medication assessment, IP dispensing. • Visit 1 (Month 1 (M1) - D30 ± 3): Following items will be recorded: treatment compliance, vital signs, blood chemistry, ECG, adverse events (AEs), concomitant medication; dispensing of new IP doses and collecting of dispensed IP at the last visit. • Visit 2 (Month 2 (M2) - D60 ± 3): Following items will be recorded: treatment compliance, AEs, concomitant medication; dispensing of new IP doses and collecting of dispensed IP at the last visit. • Visit 3 (Month 3 (M3) - D90 ± 3): Following items will be recorded: vital signs, laboratory tests (hematology, blood chemistry, electrolytes, Qmax, urinalysis, 12-lead ECG, total PSA level), concomitant medication, SFQ score, AE assessment, collecting of dispensed IP at the last visit and dispensing of new IP doses. • Visit 4 (Month 4.5 (M4) - D135 ± 3): Following items will be recorded: treatment compliance, vital signs, AEs, concomitant medication; dispensing of new IP doses and collecting of dispensed IP at the last visit. Visit 5 (Month 6 (M6)- D180 ± 3): Following items will be recorded: treatment compliance, vital signs, prostate symptom score according to IPSS, laboratory tests (hematology, blood chemistry, electrolytes, Qmax, urinalysis, 12-lead ECG, total PSA level, free-to-total PSA ratio, TRUS; concomitant medication, SFQ score, AE assessment, collecting of the previous dispensed IPs . Follow-up Phone Call (Month 7 (M7)- D210 ± 3): To record any possible AE that may occur after discontinuation of study treatment.

ELIGIBILITY:
Inclusion Criteria:

Male, age ≥ 50 years. Clinical diagnosis of benign prostate hypertrophy (BPH) . International Prostate Symptom Score (IPSS) ≥ 12 Prostate volume ≥30 ml (transrectal ultrasonography). Total serum prostate specific antigen (PSA) ≥1.5 ng/mL and ≤10 ng/mL. Free-to-total PSA ratio > 20% Maximum flow rate (Qmax) >5 mL/sec and ≤15 mL/sec and post-void residual volume of < 150 mL Willing and able to give written informed consent and comply with study procedures throughout study Able to swallow and retain oral medication Able to express personal thought and feeling Ability to read and comprehend information on the Sexual Function Inventory

Exclusion Criteria:

History or evidence of prostate cancer (e.g. positive biopsy or ultrasound, suspicious digital rectal examination).

Previous prostatic surgery (TURP, balloon dilatation, thermotherapy and stent replacement) or other invasive procedures to treat BPH.

History of flexible/rigid cystoscopy or other instrumentation of the urethra within past 7 days History of acute urine retention (AUR) within past 3 months. Any causes other than BPH result in urinary symptoms or changes in flow rate (e.g. neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute or chronic prostatitis, acute or chronic urinary tract infections).

History of breast cancer or clinical finding suggestive of malignancy. Use of any 5-alpha-reductase inhibitor (e.g. Proscar®, Propecia®), drugs with antiandrogenic properties (e.g. spironolactone, flutamide, bicalutamide, cimetidine, ketoconazole, progestational agents), drugs which induce gynecomastia or drugs which affect prostate volume, within past 6 months and throughout the study (other than as study medication). Do not use dutasteride within past 12 months. Do not use metronidazole for a long time.

Concurrent use of anabolic steroids (eg. Durabolin®). Use of phytotherapy (eg: Tadenan®, Permixon®, etc) for BPH within 2 weeks of screening visit and/or predicted to need phytotherapy during the study.

Use of any alpha-adrenoreceptor blockers (i.e. indoramin, prazosin, terazosin, tamsulosin, alfuzosin and doxazosin) within 2 weeks of screening visit and/or predicted to need any alpha blockers other than tamsulosin during the study.

Use of any alpha-adrenoreceptor agonists (e.g. pseudoephedrine, phenylephrine, ephedrine) or anticholinergics (e.g. oxybutynin, propantheline) or cholinergics (e.g. bethanecol chloride) within 48 hours prior to all uroflowmetry assessments.

Hypersensitivity to any alpha-/beta-adrenoreceptor blocker or 5-alpha-reductase inhibitor, or other chemically-related drugs.

Concurrent use of drugs known or thought to have an interaction with tamsulosin and dutasteride.

History of hepatic impairment or abnormal liver function tests at screening (defined ALT, AST, and/or alkaline phosphatase >2 times the upper limit of normal, or total bilirubin >1.5 times the upper limit of normal).

History of renal insufficiency, or serum creatinine >1.5 times the upper limit of normal at screening.

History of malignancies other than basal cell carcinoma or squamous cell carcinoma of the skin within the past 5 years. Subjects with a prior malignancy who have had no evidence of disease for at least 5 years prior to screening are eligible.

Any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within past 6 months; medically uncontrollable diabetes or peptic ulcer disease History of postural hypotension, dizziness, vertigo or any signs and symptoms of orthostasis, which in judgments of investigator, could be exacerbated by tamsulosin History of unsuccessful treatment with tamsulosin or 'first dose' hypotensive episode on initiation of alpha-1-adrenoreceptor antagonist therapy.

History of unsuccessful treatment with finasteride or dutasteride. Willing to have a child during the treatment period or within 6 months thereafter Having female partner who is a pregnant woman or in child-bearing age and refuse to use condom for sexual protection Willing to donate blood during treatment period or within 6 months thereafter. History or current evidence of drug or alcohol abuse within past 12 months. History of any illness might confound the results of the study or poses additional risk to the patient.

Participation in investigational or marketed drug trial within 30 days preceding the screening visit and/or during the study treatment

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-06-29 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants with benign prostatic hyperplasia (BPH) entered into a 6-month enrollment period followed by a6-month treatment period and a one-month follow-up period. The total duration of the study was 13 months.
Groups:
- Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg: Participants received a combination of 0.5 mg dutasteride and 0.4 mg tamsulosin capsule orally approximately 30 minutes after a meal once daily for 6 months during the treatment period. Participants were followed up to 30 days after the last dose of study medication to evaluate the safety profile of study drug.
Period: Overall Study
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Started | 59
Completed | 52
Not Completed | 7
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 59
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any On-treatment Adverse Events (AEs) or Any Serious Adverse Event (SAEs) and Treatment-related AEs
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product at any dose, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is an important medical event that jeopardizes the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, and is associated with liver injury and impaired liver function.
Time Frame: From start of study medication until follow-up (up to 7 months)
Population: Intention-to-Treat (ITT) Population: all enrolled participants regardless of whether or not study treatment was administered.
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 59
Participants
  Any AE | 13
  Any SAE | 1
  Any treatment-related AE | 3

2. Primary Outcome: Number of Participants With Any Post-treatment Adverse Events (AEs) or Any Serious Adverse Event (SAEs) and Treatment-related AEs
Description: as for outcome 1
Time Frame: From start of study medication until follow-up (up to 7 months)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 59
Participants
  Any AE | 2
  Any SAE | 1
  Any treatment-related AE | 1

3. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings at the Indicated Time Points
Description: A 12 lead ECG was measured at Screening, Month 1 (Visit 1), Month 3 (Visit 3) and Month 6 (Visit 5).
Time Frame: Screening, Month 1, Month 3 and Month 6
Population: ITT Population. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 59
Participants
  Screening, n=59 | 49
  Month 1, n=56 | 47
  Month 3, n=53 | 50
  Month 6, n=52 | 44

4. Primary Outcome: Number of Participants With Clinical Chemistry Values Shift From Normal at Baseline to Abnormal at Any Time Post-Baseline
Description: Blood samples were collected at Screening, Month 1 (Visit 1), Month 3 (Visit 3) and Month 6 (Visit 5) for chemistry laboratory assessments. Clinical chemistry parameters included alanine aminotrasferase (ALT), aspartate aminotrasferase (AST), creatinine, glucose, potassium, protein, sodium and urea. The number of participants with a shift from normal at Baseline to abnormal at any time post-Baseline for a clinical chemistry parameter are summarized.
Time Frame: Screening, Month 1, Month 3 and Month 6
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 56
Participants
  ALT, n=48 | 9
  AST, n=49 | 6
  Creatinine, n=51 | 9
  Glucose, n=47 | 8
  Potassium, n=52 | 1
  Protein, n=56 | 4
  Sodium, n=53 | 0
  Urea, n=54 | 7

5. Primary Outcome: Number of Participants With Hematology Values Shift From Normal at Baseline to Abnormal at Any Time Post-Baseline
Description: Blood samples were collected at Screening, Month 3 (Visit 3) and Month 6 (Visit 5) for hematology laboratory assessments. Hematology parameters included basophils, leukocytes, hemoglobin (HGB), eosinophils, erythrocytes (ery), ery mean Corpuscular HGB concentration, ery mean corpuscular HGB, ery distribution width, lymphocytes, hematocrit, monocytes, neutrophils and platelets. The number of participants with a shift from normal at Baseline to abnormal at any time post-Baseline for hematology parameters are summarized.
Time Frame: Screening, Month 3 and Month 6
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 56
Participants
  Basophils/Leukocytes, n=54 | 0
  Eosinophils/Leukocytes, n=46 | 5
  Ery Mean Corpuscular HGB Concentration, n=44 | 22
  Ery Mean Corpuscular Hemoglobin, n=36 | 6
  Ery Mean Corpuscular Volume, n=42 | 4
  Erythrocytes, n=49 | 3
  Erythrocytes Distribution Width, n=4 | 3
  Hematocrit, n=48 | 7
  Hemoglobin, n=49 | 2
  Leukocytes, n=47 | 7
  Lymphocytes/Leukocytes, n=53 | 1
  Monocytes/Leukocytes, n=52 | 1
  Neutrophils/Leukocytes, n=41 | 5
  Platelets, n=53 | 1

6. Primary Outcome: Number Participants With a Negative or Positive Response at the Indicated Time Points
Description: Urine samples were collected at Screening (SC), Month 3 (3M) and Month 6 (6M) for urinalysis laboratory assesment. Final value (FV) is defined as the latest post-Baseline value available in the study for each parameter.Urinalysis parameters included erythrocytes, glucose, ketones, leukocytes and protein. Number of participants with a negative (NEG) or positive (POS) response at the indicated time points are summarized.
Time Frame: Screening, Month 3 and Month 6
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 59
Participants
  Erythrocytes, SC, POS, n=59 | 4
  Erythrocytes, SC, NEG, n=59 | 55
  Erythrocytes, 3M, POS, n=54 | 6
  Erythrocytes, 3M, NEG, n=54 | 48
  Erythrocytes, 6M, POS, n=52 | 6
  Erythrocytes, 6M, NEG, n=52 | 46
  Erythrocytes, FV, POS, n=54 | 7
  Erythrocytes, FV, NEG, n=54 | 47
  Glucose, SC, POS, n=59 | 3
  Glucose, SC, NEG, n=59 | 56
  Glucose, 3M, POS, n=54 | 1
  Glucose, 3M, NEG, n=54 | 53
  Glucose, 6M, POS, n=52 | 0
  Glucose, 6M, NEG, n=52 | 52
  Glucose, FV, POS, n=54 | 0
  Glucose, FV, NEG, n=54 | 54
  Ketones, SC, POS, n=59 | 0
  Ketones, SC, NEG, n=59 | 59
  Ketones, 3M, POS, n=54 | 2
  Ketones, 3M, NEG, n=54 | 52
  Ketones, 6M, POS, n=52 | 1
  Ketones, 6M, NEG, n=52 | 51
  Ketones, FV, POS, n=54 | 1
  Ketones, FV, NEG, n=54 | 53
  Leukocytes, SC, POS, n=59 | 3
  Leukocytes, SC, NEG, n=59 | 56
  Leukocytes, 3M, POS, n=54 | 0
  Leukocytes, 3M, NEG, n=54 | 54
  Leukocytes, 6M, POS, n=52 | 6
  Leukocytes, 6M, NEG, n=52 | 46
  Leukocytes, FV, POS, n=54 | 6
  Leukocytes, FV, NEG, n=54 | 48
  Protein, SC, POS, n=59 | 9
  Protein, SC, NEG, n=59 | 50
  Protein, 3M, POS, n=54 | 6
  Protein, 3M, NEG, n=54 | 48
  Protein, 6M, POS, n=52 | 7
  Protein, 6M, NEG, N=52 | 45
  Protein, FV, POS, n=54 | 8
  Protein, FV, NEG, n=54 | 46

7. Primary Outcome: Change From Baseline in Total Prostate -Specific Antigen (PSA) at the Indicated Time Points
Description: Serum sample was collected at Baseline, Month 3 and Month 6 for assesment of total PSA. PSA is a substance produced by prostate gland, and the elevated level of PSA indicates prostate cancer or any other non-cancerous condition related to prostate. Change from Baseline in total PSA at Month 3 and Month 6 was calculated as value at specified visist minus Baseline value.
Time Frame: Baseline, Month 3 and Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Microgram per liter (ug/L)
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 54
Microgram per liter (ug/L)
  Month 3, n=54 | -1.499 (1.2263)
  Month 6, n=52 | -1.824 (1.2413)

8. Primary Outcome: Free to Total PSA Ratio at the Indicated Time Points
Description: Serum sample was collected at Screening (Baseline for participants with Free to Total PSA ratio at Month 6), and Month 6 for assessment of free to total PSA ratio. PSA is a substance produced by prostate gland, and the elevated level of PSA indicates prostate cancer or any other non-cancerous condition related to prostate. Free to total PSA ratio at Baseline for participants with free to total PSA Ratio at Month 6 and free to total PSA ratio at month 6 are presented.
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 57
Ratio
  Baseline, n=50 | 28.207 (10.5868)
  Month 6, n=52 | 24.887 (8.1112)

9. Secondary Outcome: Change From Baseline in the International Prostate Symptom Score (IPSS) at Month 6
Description: The IPSS is a screening tool used to assess the symptoms of prostate related disease. The IPSS questionnaire consists of seven symptoms questions including feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia, each referring to during the last month, and each involving assignment of a score from 0 to 5 (no symptoms to almost always symptoms) for a total of maximum 35 points. IPSS total is the sum of the scores of seven questions; therefore, the possible total score ranges from 0 to 35 (0-7: Mildly symptomatic; 8-19: Moderately symptomatic; 20-35: Severely symptomatic). IPSS was assessed at Baseline and Month 6. Change from Baseline was calculated as Month 6 IPSS score- minus Baseline IPSS score.
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 52
Scores on a scale | -8.3 (3.92)
Statistical Analysis 1: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

10. Secondary Outcome: Change From Baseline in Maximum Rate of Urinary Flow (Qmax) at the Indicated Time Points
Description: The Qmax is used as an indicator for the diagnosis of enlarged prostate. A lower Qmax may indicate that the enlarged prostate. Qmax was assessed at Baseline (screening), Month 3 and Month 6. Change from Baseline was calculated as Qmax score at specified timepoint minus the Baseline Qmax score.
Time Frame: Baseline, Month 3 and Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Mililiter/seconds
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Number analyzed (Participants) | 54
Mililiter/seconds
  Month 3, n=54 | 2.77 (4.361)
  Month 6, n=52 | 2.01 (3.684)
Statistical Analysis 1: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — for Month 3
Statistical Analysis 2: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — for Month 6

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until follow-up (up to Month 7).
Description: SAEs and non-serious AEs were collected for the participants of the ITT population, comprised of all enrolled participants regardless of whether or not study treatment was administered.
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg
Serious Adverse Events (participants affected / at risk) | 1/59
Other Adverse Events (participants affected / at risk) | 0/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg (N=59)
Hepatic Enzyme Increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.